CLINICAL TRIAL: NCT01524913
Title: A Double Blind Randomised Study Comparing Hyaluronic Acid, Corticosteroid and Placebo During Arthrocentesis for Temporomandibular Joint Dysfunction
Brief Title: A Double Blind Study Comparing Hyaluronic Acid, Corticosteroid and Placebo During Arthrocentesis for Temporomandibular Joint (TMJ) Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: University of California, Los Angeles (Other); Oregon Health and Science University (Other); University of Minnesota (Other); University of Cincinnati (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Gary F Bouloux MD, DDS, MDSc, FRACDS, FRACDS, National PI, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00018682; Arthrocentesis (Other: Other)
Record Dates: First submitted 2012-01-29; First posted 2012-02-02 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Temporomandibular Joint Dysfunction; Pain; Arthrocentesis
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain | interventions — Hyaluronic Acid; Adrenal Cortex Hormones; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hyaluronic acid (Experimental)
  Interventions: Drug: Hyaluronic acid
- Corticosteroid (Active Comparator)
  Interventions: Drug: Corticosteroid
- Saline (Placebo Comparator)
  Interventions: Drug: Lactated Ringers

INTERVENTIONS:
Drug: Hyaluronic acid — 1 cc hyalgan to be injected into superior joint space
  Arms: Hyaluronic acid
Drug: Corticosteroid — 1cc celestone (6 mg/cc) will be injected into the joint space
  Arms: Corticosteroid
Drug: Lactated Ringers — 1 cc lactated ringers solution will be injected into the joint space
  Arms: Saline

SUMMARY:
The purpose of this study is to determine whether the administration of hyaluronic acid or corticosteroid during arthrocentesis of the temporomandibular joint provides additional pain relief and improved function.

The overall hypothesis for the study is that hyalgan will result in a 30% reduction in the mean visual analogue scale (VAS) at one month when compared to celestone and placebo.

DETAILED DESCRIPTION:
This study will enroll patients with temporomandibular joint dysfunction who are deemed appropriate candidates for irrigation of their jaw joints secondary to pain or limited opening. At the completion of the joint irrigation subjects will be injected by one of three different products to determine if the additional injection results in a further decrease in jaw joint pain and improved opening. Subjects will be followed for 3 months. Those who do not show improvement may be candidates for additional treatment.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years
* arthralgia of one or both temporomandibular joints
* Wilkes II to IV internal derangement of the symptomatic joint OR
* limited opening of <35 mm

Exclusion Criteria:

* myofascial pain as the primary source of pain

  * cervical pain as the primary source of pain
* systemic arthropathy
* fibromyalgia
* use of NSAIDS within 48 hours
* allergy to study medications
* edentulous subjects
* pregnancy or breast feeding
* current physical therapy, muscle relaxants or antiseizure medications
* current use of a splint issued within last 12 weeks

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary F Bouloux, MD, DDS, Principal Investigator — Emory University
Locations (5):
- United States (5):
  - University California Los Angeles, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - University of Cinncinati, Cinncinati, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Bouloux GF, Chou J, Krishnan D, Aghaloo T, Kahenasa N, Smith JA, Giannakopoulos H. Is Hyaluronic Acid or Corticosteroid Superior to Lactated Ringer Solution in the Short-Term Reduction of Temporomandibular Joint Pain After Arthrocentesis? Part 1. J Oral Maxillofac Surg. 2017 Jan;75(1):52-62. doi: 10.1016/j.joms.2016.08.006. Epub 2016 Aug 20. PMID 27632069
- [Result] Bouloux GF, Chou J, Krishnan D, Aghaloo T, Kahenasa N, Smith JA, Giannakopoulos H. Is Hyaluronic Acid or Corticosteroid Superior to Lactated Ringer Solution in the Short Term for Improving Function and Quality of Life After Arthrocentesis? Part 2. J Oral Maxillofac Surg. 2017 Jan;75(1):63-72. doi: 10.1016/j.joms.2016.08.008. Epub 2016 Aug 20. PMID 27632067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from patients referred to the oral and maxillary surgery services at Emory University, the University of Pennsylvania, the University of California - Los Angeles, the University of Cincinnati, and the Oregon Health Science University. All patients were referred for management of temporomandibular joint (TMJ) pain.
Pre-assignment Details: A total of 105 patients were screened; three did not meet inclusion and exclusion criteria, resulting in 102 participants who were randomized and began the study treatment.
Groups:
- Corticosteroid: Participants in this group received 1 milliliter (mL) of Celestone (6mg/mL) injected into the the superior joint space.
- Hyaluronic Acid: Participants in the group received 1milliliter (mL) of Hyalgan (10 mg/mL) injected into the superior joint space.
- Saline Placebo: Participants in this group received 1 milliliter (mL) of lactated Ringer's solution injected into the superior joint space.
Period: Overall Study
Arm/Group | Corticosteroid | Hyaluronic Acid | Saline Placebo
Started | 35 | 36 | 31
Completed | 31 | 36 | 31
Not Completed | 4 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population includes all participants who met eligibility criteria, were randomized to a study arm, and received their assigned study treatment.
Groups:
- Corticosteroid: Participants in this group received 1mL of Celestone (6mg/mL) injected into the the superior joint space.
- Hyaluronic Acid: Participants in the group received 1mL of Hyalgan (10 mg/mL) injected into the superior joint space.
- Saline Placebo: Participants in this group received 1mL of lactated Ringer's solution injected into the superior joint space.
- Total: Total of all reporting groups
Arm/Group | Corticosteroid | Hyaluronic Acid | Saline Placebo | Total
Number analyzed (Participants) | 35 | 36 | 31 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (18.4) | 44.3 (17.2) | 51.8 (17.2) | 45.0 (18.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 28 | 89
  Male | 4 | 6 | 3 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 6 | 7 | 6 | 19
  White | 25 | 28 | 23 | 76
  Asian | 1 | 0 | 1 | 2
  Other | 3 | 1 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 35 | 36 | 31 | 102
Headache [Count of Participants; unit: Participants]
  Yes | 19 | 17 | 16 | 52
  No | 16 | 19 | 15 | 50
Migraine [Count of Participants; unit: Participants]
  Yes | 12 | 9 | 7 | 28
  No | 23 | 27 | 24 | 74
Prior TMJ Surgery [Count of Participants; unit: Participants]
  Yes | 5 | 4 | 1 | 10
  No | 30 | 32 | 30 | 92
Capsular Pain [Count of Participants; unit: Participants]
  Yes | 26 | 28 | 24 | 78
  No | 9 | 8 | 7 | 24
Myofascial Pain [Count of Participants; unit: Participants]
  Yes | 15 | 24 | 20 | 59
  No | 20 | 12 | 11 | 43
Cervical Pain [Count of Participants; unit: Participants]
  Yes | 11 | 13 | 9 | 33
  No | 24 | 23 | 22 | 69
Clicking Jaw [Count of Participants; unit: Participants]
  Yes | 14 | 14 | 9 | 37
  No | 21 | 22 | 22 | 65
Crepitus [Count of Participants; unit: Participants]
  Yes | 5 | 6 | 2 | 13
  No | 30 | 30 | 29 | 89

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Between Baseline and Month 1 Scores
Description: The change in pain level was assessed using a single-item visual analogue pain scale at Baseline (preoperatively) and at Month 1. Participants indicate their level on pain on a scale of 0 (no pain) to 10 (worst pain imaginable). The right and left side of each participant's jaw was evaluated separately. The change in pain score was obtained by subtracting the Month 1 score from the Baseline score and a negative value indicates a reduction in pain level.
Time Frame: Baseline (preoperation), Month 1
Population: The population at this time point consists of study participants who received their assigned intervention and were not lost to follow up by the Month 1 assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Corticosteroid | Hyaluronic Acid | Saline Placebo
Number analyzed (Participants) | 31 | 36 | 31
units on a scale
  Change in Pain - Right Side | -1.1 (2.8) | -1.7 (3.0) | -2.6 (2.8)
  Change in Pain - Left Side | -2.0 (3.1) | -2.1 (3.1) | -2.3 (3.2)

2. Secondary Outcome: Change in Maximum Incisal Opening (MIO) Between Baseline, Month 1, and Month 3
Description: Range of motion was assessed at Baseline (preoperatively) and again at Months 1 and 3 using a millimeter ruler for maximum incisal opening. MIO was measurements were taken for maximum opening without and with pain.
Time Frame: Baseline (preoperation), Month 1, Month 3
Population: The population for MIO analysis consists of participants having a measurement at each specified time point. The decline in the number of participants over time is due to participants who were lost to follow-up as the study progressed and one participant who attended the Month 3 visit but did not provide data for the MIO assessment.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Corticosteroid | Hyaluronic Acid | Saline Placebo
Number analyzed (Participants) | 35 | 36 | 31
millimeters
  Baseline MIO without pain | 28.3 (8.4) | 27.9 (11.2) | 25.7 (7.5)
  Baseline MIO maximum | 37.0 (8.5) | 33.9 (10.3) | 34.1 (7.8)
  Month 1 MIO without pain: number analyzed (Participants) | 31 | 36 | 31
  Month 1 MIO without pain | 35.0 (9.4) | 31.7 (11.4) | 29.6 (10.6)
  Month 1 MIO maximum: number analyzed (Participants) | 31 | 36 | 31
  Month 1 MIO maximum | 39.0 (10.5) | 36.8 (11.2) | 37.4 (6.7)
  Month 3 MIO without pain: number analyzed (Participants) | 19 | 17 | 15
  Month 3 MIO without pain | 36.1 (11.3) | 33.9 (11.7) | 35.7 (5.0)
  Month 3 MIO maximum: number analyzed (Participants) | 19 | 17 | 15
  Month 3 MIO maximum | 37.8 (15.0) | 38.3 (13.2) | 39.3 (5.3)

3. Secondary Outcome: Jaw Function Limitation Scale (JFLS) Score
Description: The Jaw Function Limitation Scale (JFLS) is an 8 item survey where respondents indicate the presence or absence of problems with chewing, drinking, eating hard food, eating soft food, smiling or laughing, yawning, swallowing, and talking. Responses of "no" are scored as "0" and responses of "yes" are scored as "1". The total score categorizes jaw limitation as: none (0), mild (1-3), moderate (4-6), and severe (7-8).
Time Frame: Month 1
Population: The population at this time point consists of study participants who received the intervention they were randomized to and were not lost to follow-up before the Month 1 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Corticosteroid | Hyaluronic Acid | Saline Placebo
Number analyzed (Participants) | 31 | 36 | 31
Participants
  None | 3 | 5 | 6
  Mild | 18 | 14 | 14
  Moderate | 9 | 14 | 9
  Severe | 1 | 3 | 2

4. Secondary Outcome: Jaw Function Limitation Scale (JFLS) Score
Description: as for outcome 3
Time Frame: Month 3
Population: The population at this time point consists of study participants who received the intervention they were randomized to, were not lost to follow-up before the Month 3 visit, and completed assessments at the Month 3 visit (one participant did not provide JFLS data at the Month 3 time point).
Measure: Count of Participants; unit: Participants
Arm/Group | Corticosteroid | Hyaluronic Acid | Saline Placebo
Number analyzed (Participants) | 19 | 17 | 15
Participants
  None | 5 | 5 | 6
  Mild | 8 | 7 | 5
  Moderate | 5 | 4 | 4
  Severe | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed up to three months after arthrocentesis. Allergic reactions were watched for during the procedure and during the 30 minute recovery period after the procedure. Post injection flare was monitored after 1 month. All other adverse events were monitored during for three months post-procedure.
Description: Adverse events were actively sought, including allergic reactions (anaphylaxis, angioedema, urticaria), post-injection flare, hospital admission, the need for additional procedures to prevent or limit permanent injury, and death and other life threatening events. Given the extensive safe track record of hyaluronic acid and the corticosteroid Celestone, no adverse events were expected to occur.
Arm/Group | Corticosteroid | Hyaluronic Acid | Saline Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/31
Other Adverse Events (participants affected / at risk) | 0/35 | 0/36 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes